CLINICAL TRIAL: NCT01070355
Title: The Effects of Eicosapentaenoic Acid (EPA) on Biomarkers of Growth and Vascularity in Human Colorectal Cancer Liver Metastases (The EPA for Metastasis Trial)
Brief Title: Eicosapentaenoic Acid (EPA) for Treatment of Colorectal Cancer Liver Metastases
Acronym: EMT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Mark Hull, Professor, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GA09/9094; 2009-015903-22 (EudraCT Number)
Record Dates: First submitted 2010-02-12; First posted 2010-02-18 (Estimated); Last update posted 2011-10-21 (Estimated); Status verified 2011-10

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Neoplasms; Fish Oils; Fatty Acids, Omega-3; Eicosapentaenoic Acid; Liver Metastases; Randomised Controlled Trial
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 2 capsules twice daily
  Interventions: Drug: Placebo
- Eicosapentaenoic acid free fatty acid (Active Comparator): 2g daily (2 x 500mg capsules twice daily)
  Interventions: Drug: Eicosapentaenoic acid free fatty acid

INTERVENTIONS:
Drug: Eicosapentaenoic acid free fatty acid — An enteric-coated preparation of 99% pure omega-3 polyunsaturated fatty acid (PUFA) eicosapentaenoic acid as the free fatty acid. 500mg capsules, 2 taken twice daily for 2-6 weeks before liver resection.
  Other Names: ALFA
  Arms: Eicosapentaenoic acid free fatty acid
Drug: Placebo — 2 capsules taken twice daily for 2-6 weeks before liver resection.
  Arms: Placebo

SUMMARY:
Eicosapentaenoic acid (EPA) is a naturally occuring omega-3 polyunsaturated fatty acid found in oily fish. EPA has anti-colorectal (bowel) cancer activity in experimental models. This trial will test whether EPA reduces markers of tumour growth, and is safe and well tolerated,in patients with colorectal cancer liver metastases awaiting surgery.

DETAILED DESCRIPTION:
A double-blind, randomised, placebo-controlled trial of eicosapentaenoic acid (EPA), in the free fatty acid form, 2g daily in patients who will undergo liver resection surgery for colorectal cancer liver metastases.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Either sex
* Liver resection deemed clinically appropriate for management of metastatic colorectal cancer
* Duration between decision to perform liver resection and surgery greater than 2 weeks
* Ability to give written informed consent and follow study protocol
* Telephone contact possible

Exclusion Criteria:

* Neo-adjuvant chemotherapy for colorectal cancer (CRC) liver metastasis
* Chemotherapy for any cancer in the previous 3 months
* Known bleeding diathesis or anticoagulation therapy
* Fish or seafood allergy
* Use of fish oil supplements (eg. cod liver oil) and unwilling to stop for the duration of the study
* Pregnancy
* Non-aspirin non-steroidal anti-inflammatory (NSAID) or corticosteroid use
* Renal impairment (serum creatinine >150)
* Active inflammatory disease (e.g. Inflammatory Bowel Disease, Rheumatoid Arthritis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2010-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Histological Ki67 cancer cell proliferation index | at surgery 2-6 weeks after randomisation

SECONDARY OUTCOMES:
Histological neo-CK18 cancer cell apoptosis index | at surgery 2-6 weeks after randomisation
Histological tumour CD31-positive cell microvessel density | at surgery 2-6 weeks after randomisation
Safety and tolerability of EPA treatment | Every 2 weeks whilst patient is taking study medication
Metastatic tissue and healthy liver tissue fatty acid composition and prostaglandin levels | at surgery 2-6 weeks after randomisation
Plasma markers of prostaglandin metabolism | 1. Baseline 2. after approx 4 weeks of study medication (immediately prior to surgery). 3. Six weeks after liver resection (no study medication)
Platelet aggregation | 1. Baseline 2. after approx 4 weeks of study medication (immediately prior to surgery). 3. Six weeks after liver resection (no study medication)
Urinary markers of prostaglandin metabolism | 1. Baseline 2. after 2 weeks of study medication 3. after approx 4 weeks of study medication (immediately prior to surgery). 4. Six weeks after liver resection (no study medication)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Hull, PhD, FRCP, Principal Investigator — Leeds Institute of Molecular Medicine, University of Leeds
Locations (1):
- Leeds Institute of Molecular Medicine, St James's University Hospital, Leeds, West Yorkshire, United Kingdom

REFERENCES:
- [Derived] Cockbain AJ, Volpato M, Race AD, Munarini A, Fazio C, Belluzzi A, Loadman PM, Toogood GJ, Hull MA. Anticolorectal cancer activity of the omega-3 polyunsaturated fatty acid eicosapentaenoic acid. Gut. 2014 Nov;63(11):1760-8. doi: 10.1136/gutjnl-2013-306445. Epub 2014 Jan 27. PMID 24470281